CLINICAL TRIAL: NCT01065363
Title: Project of Health Promotion and Management for Hepatitis B Carriers in NTU Campus
Brief Title: Health Promotion and Management for Hepatitis B Carriers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Jin-Shin Lai/ Attending physician, Department of physical medicine and rehabilitation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200906036R
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B virus DNA; Metabolic factor; Body mass index; Obesity; Insulin resistance; Lifestyle factor; Preventive Medicine; Health Promotion
MeSH Terms: conditions — Hepatitis B, Chronic; Obesity; Insulin Resistance | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle conseling (Experimental)
  Interventions: Behavioral: standardized exercise program and dietary counseling

INTERVENTIONS:
Behavioral: standardized exercise program and dietary counseling — Lecture, 12 weeks Standardized exercise program, 12 weeks Dietary counseling, 12 weeks Information platform, 12 weeks

SUMMARY:
The investigators propose a project of preventive medicine with concern of local context in Taiwan. The target population includes all staff and faculty members, students, and alumni of a university in Northern Taiwan, with chronic hepatitis B infection. The intervention of this project includes standardized lectures, sports courses, nutrition courses, and an information platform. The investigators will evaluate the efficacy after the intervention, like the reduction of hepatitis B viral load and the associated anthropometric parameters. The results of this project will be initially served as a pilot study for this cohort, and applicated as a promising basis for health promotion.

ELIGIBILITY:
Inclusion Criteria:

* Participants were recruited from students, alumni, faculty and staff members with chronic HBV infection (positive HBsAg serostatus ≥6 months) in a university of northern Taiwan from August 1, 2009 to July 01, 2010. Only participants aged 18 and older were included.

Exclusion Criteria:

* Excluded were:

  * (a) those who had been diagnosed as chronic liver diseases like chronic hepatitis C infection (Anti-HCV (+)), autoimmune hepatitis, Wilson disease, alcoholic liver diseases, drug-related hepatitis, decompensated liver diseases, cirrhosis, or malignant hepatic tumors;
* (b) those who had undergone liver transplantation or major operations for liver except cholecystectomy;
* (c) men who consumed more than 30 gram of alcohol per week or women who consumed more than 20 gram of alcohol per week;
* (d) women who were pregnant;
* (e) those who had current medications for any types of chronic diseases except for hyperglycemia, elevated blood pressure, or dyslipidemia within six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of relative serum HBV DNA levels | three months

SECONDARY OUTCOMES:
anthropometric index | three months

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shin Lai, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation
Locations (1):
- National Taiwan University Health Center, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://ann.cc.ntu.edu.tw/asp/ShowContent.asp?num=16309